CLINICAL TRIAL: NCT06221579
Title: An Intergenerational, Cognitively Enriched Lifestyle Intervention for Patients With a Mild Cognitive Impairment (MCI) and Their Children.
Brief Title: An Intergenerational, Cognitively Enriched Intervention for MCI Patients and Their Children.
Acronym: MCI-project
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCI-project - ONZ-2023-0246
Record Dates: First submitted 2023-12-06; First posted 2024-01-24 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: Interviews with MCI patients to develop the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interview (Experimental): Conducting interviews with MCI patients to identify their needs and preferences related to the intervention to be developed
  Interventions: Other: No intervention, interviews with MCI patients as part of the development phase

INTERVENTIONS:
Other: No intervention, interviews with MCI patients as part of the development phase — No intervention, interviews with MCI patients as part of the development phase

SUMMARY:
In 2018, approximately 50 million people received a diagnosis of dementia, which is projected to triple by 2050. To mitigate the increase in dementia, it is crucial to prevent cognitive decline in at risk groups, such as older adults with mild cognitive impairment (MCI). Recent research has demonstrated that combining physical (PA) and cognitive activities yields positive effects on the cognitive health of older adults. However, it is essential to explore effective ways of implementing this approach for MCI patients as it may help prevent dementia. An intergenerational program offers a novel and innovative method to achieve this goal by involving both older and younger generations in a single (exercise) program aimed at promoting the health behavior of both groups. Engaging children in an intergenerational, cognitively enriched exercise program for MCI patients primarily benefits the older adults while also providing advantages for the adult children. Therefore, this intergenerational project serves as a valuable and motivating force to enhance the physical, cognitive, and psychosocial health of MCI patients, with a secondary aim of positively impacting the adult children.

Phase 1 of this project (=current study) involves developing the intergenerational, cognitively enriched exercise program. This will be accomplished using a theoretical framework in combination with a co-creation approach, which actively involves MCI patients in the intervention development. Ten thinkaloud interviews (lasting approximately 2 hours) will be conducted with MCI patients and one of their adult children. The insights gained from these interviews will be used to adapt an existing exercise intervention for MCI patients according to their specific needs. Prior to the interview, participants will also be asked to complete a short questionnaire that collects basic demographic information.

DETAILED DESCRIPTION:
In 2018, approximately 50 million people received a diagnosis of dementia, which is projected to triple by 2050. To mitigate the increase in dementia, it is crucial to prevent cognitive decline in at risk groups, such as older adults with mild cognitive impairment (MCI). Recent research has demonstrated that combining physical (PA) and cognitive activities yields positive effects on the cognitive health of older adults. However, it is essential to explore effective ways of implementing this approach for MCI patients as it may help prevent dementia.

An intergenerational program offers a novel and innovative method to achieve this goal by involving both older and younger generations in a single (exercise) program aimed at promoting the health behavior of both groups. Engaging children in an intergenerational, cognitively enriched exercise program for MCI patients primarily benefits the older adults while also providing advantages for the adult children. Therefore, this intergenerational project serves as a valuable and motivating force to enhance the physical, cognitive, and psychosocial health of MCI patients, with a secondary aim of positively impacting the adult children.

Phase 1 of this project (=current study) involves developing the intergenerational, cognitively enriched exercise program. This will be accomplished using a theoretical framework in combination with a co-creation approach, which actively involves MCI patients in the intervention development. Ten thinkaloud interviews (lasting approximately 2 hours) will be conducted with MCI patients and one of their adult children. The insights gained from these interviews will be used to adapt an existing exercise intervention for MCI patients according to their specific needs. Prior to the interview, participants will also be asked to complete a short questionnaire that collects basic demographic information.

ELIGIBILITY:
Inclusion criteria:

1. MCI Diagnosis: Individuals with mild cognitive impairment (MCI) are eligible to participate, without a formal dementia diagnosis.
2. MCI Type: Both amnestic and non-amnestic MCI individuals qualify for participation.
3. Adult Child: Must have an adult child willing to participate in the program, free from serious health issues, both physically and cognitively.

Exclusion criteria:

1. Dementia Diagnosis: Individuals formally diagnosed with dementia cannot participate.
2. MCI from Specific Causes: Excludes those with MCI caused by frontotemporal dementia or Parkinson's.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Needs Assessment in MCI Patients and Their Children based on Think Aloud Interviews | 2 hours
  The interviews utilized a guide with "needs assessment cards" based on literature findings, addressing difficulties, motivators, and specific needs of MCI patients and their children. Participants were encouraged to use cards for relevance but had the freedom to express additional difficulties or motivators. Instructions provided clarity at the beginning of the card bundle. Collected data will be aggregated by categorizing responses from 'needs assessment cards' into themes, providing insights into common challenges, motivators, and specific needs. This streamlined analysis aids in identifying patterns and tailoring interventions for MCI patients and their children.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vanlangenhove, Dr., Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No